CLINICAL TRIAL: NCT04183738
Title: The Impact of Co-infections on Inflammation in Patients Commencing Second-line Antiretroviral Therapy. A Sub-study of D²EFT (Dolutegravir and Darunavir Evaluation in Adults Failing Therapy)
Brief Title: Inflammation and Co-Infections in D²EFT
Acronym: i2-D²EFT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: In the context of COVID-19 pandemic.
Sponsor: Kirby Institute (Other Government)
Collaborators: Frederick National Laboratory for Cancer Research (Unknown); UNITAID (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); ViiV Healthcare (Industry); Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-10-i2-DEFT; 18Q065 (Other Grant/Funding Number: NIAID via Leidos)
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: HIV-infection/Aids; Human Herpesvirus 4 Infections; Cytomegalovirus Infections; Human Herpesvirus 8 Infection; Human Papilloma Virus
Keywords: HIV; IL-6; EBV; CMV; HHV8; HPV; inflammation; co-infections; opportunistic infections; AIDS and non-AIDS defining cancers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Epstein-Barr Virus Infections; Cytomegalovirus Infections; Inflammation; Coinfection; Opportunistic Infections | interventions — Nucleosides; Darunavir; Ritonavir; dolutegravir

STUDY DESIGN:
Intervention Model Description: Observational cohort nested within the parent open label phase III/IV randomised controlled trial of simplified second-line therapy, D²EFT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SOC (Active Comparator): darunavir/ritonavir 800/100mg + 2 NRTIs po od
  Interventions: Drug: NRTIs; Drug: Darunavir; Drug: Ritonavir
- DOL (Experimental): darunavir/ritonavir 800/100mg + dolutegravir 50mg po od
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Dolutegravir
- D2N (Experimental): dolutegravir 50mg + tenofovir + emtricitabine or lamivudine po od
  Interventions: Drug: NRTIs; Drug: Dolutegravir

INTERVENTIONS:
Drug: NRTIs — In SOC arm, choice of NRTIs determined by clinician, guided by either genotypic resistance testing or use of a protocol-specified algorithm for N(t)RTI selection.
  In D2N arm, NRTIs are predetermined.
  Other Names: Nucleoside/Nucleotide Reverse Transcription Inhibitors
  Arms: D2N; SOC
Drug: Darunavir — 800mg tablet by mouth once daily for 96 weeks.
  Other Names: Prezista
  Arms: DOL; SOC
Drug: Ritonavir — 100mg tablet by mouth once daily for 96 weeks.
  Other Names: Norvir
  Arms: DOL; SOC
Drug: Dolutegravir — 50mg tablet by mouth once daily for 96 weeks.
  Other Names: Tivicay
  Arms: D2N; DOL

SUMMARY:
i2-D²EFT substudy is an observational cohort nested within the parent D²EFT study (NCT03017872). D²EFT goal is to compare the standard of care second-line antiretroviral therapy in people living with HIV whose first-line non nucleoside reverse transcriptase-based regimen failed, to two simpler regimens. Approximately 1,000 participants will be enrolled in D²EFT.

Commencing a second-line ART is an important moment when the level of inflammation in participants may be elevated due to first-line ART failure; this level of inflammation should then decrease with the commencement of a new second-line treatment and would be expected to normalise by 48 weeks of second-line treatment, if successful.

The investigators propose to study other factors which can influence the decrease of inflammation. The investigators hypothesise that co-infections may play a role in persistent inflammation. The key-infections of interest will be common frequent infections encounter throughout the world: Human Herpes virus 8, Epstein-Barr virus, Cytomegalovirus and Human papillomavirus, tuberculosis, malaria and other key opportunistic infections. Possible changes of level of inflammation (using the serum level of Interleukin 6) in approximately 200 participants of the D²EFT study will be investigated and measured. The hypothesis is that the presence of other infections than HIV may influence the level of inflammation in participants in therapeutic success.

DETAILED DESCRIPTION:
i2-D²EFT substudy an observational cohort nested within the parent open label phase III/IV randomised controlled trial of simplified second-line therapy, D²EFT (NCT03017872). Participants consenting to D²EFT study will be randomised within the three arms: either ritonavir-boosted darunavir plus two nucleosides or dolutegravir plus two predetermined nucleosides (tenofovir disoproxil fumarate plus lamivudine or emtricitabine) or ritonavir-boosted darunavir plus dolutegravir. Enrolment into the i2-D²EFT substudy is voluntary and optional for participants in D²EFT. Parameters relevant to i2-D²EFT substudy including demographics, arm of randomised ART, HIV history, physical examination, immunological and virological results, episodes of co-infections and adverse events due to any infection or malignancies at required time points will be collected as part of D²EFT study. Substudy specific assessments performed at baseline and at weeks 48 include sample collection for IL-6 dosage plus EBV/CMV/HHV8 testing, and optional anal/cervical HPV screening.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the eligibility criteria for D²EFT randomisation;
* Being able to give a written informed consent for the i2-D²EFT sub-study.

Exclusion Criteria:

* Unwilling to comply with the i2-D²EFT protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-12-19 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IL-6 level at week 48 | At week 0 and week 48
  To compare the change of a biomarker of inflammation (IL-6) in participants who achieve HIV virological suppression (defined as peripheral blood viral load below 50 copies/mm3 at week 48) across the three study arms according to the presence (or not) of active key-co-infections (HHV8, EBV, CMV, HPV) at baseline and week 48, and the occurrence (or not) within these 48 weeks of any infection (co-infections or opportunistic infections).
Change from baseline of presence/absence of active key co-infections at week 48 | At week 0 and week 48
  Active key-co-infections (HHV8, EBV, CMV, HPV) at baseline and week 48, and the occurrence (or not) within these 48 weeks of any infection (co-infections or opportunistic infections).

SECONDARY OUTCOMES:
Prevalence of HHV8, EBV and CMV and of cervical and anal HPV | At week 0
  To describe the prevalence of HHV8, EBV and CMV (defined by serological assays) and of cervical and anal HPV (defined by tissue HPV deoxyribonucleic acid (DNA) detection) at baseline, in the D2EFT cohort, by geographic region, route of HIV transmission, and other demographic and disease variables.
Occurrence of active HHV8, EBV and CMV | At week 48
  To compare the occurrence of active HHV8, EBV and CMV (defined by a detectable peripheral blood viral load) in participants with and without HIV virological suppression at 48 weeks, across the three arms of D²EFT.
Change from baseline in rates of detection of cervical and anal HPV infection at week 48 | At week 0 and week 48
  To compare rates of detection of cervical and anal HPV infection (defined by tissue HPV DNA detection) between baseline and week 48 in participants with and without HIV virological suppression at 48 weeks across the three arms of D²EFT.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polizzotto, MD, PhD, Principal Investigator — Kirby Institute, UNSW Sydney, Australia

IPD SHARING:
Plan to Share IPD: No